CLINICAL TRIAL: NCT01148056
Title: A Phase II Study of Neoadjuvant Short Course Intensity Modulated Radiation Therapy (IMRT) for Patients With Rectal Cancer: An Analysis of Quality of Life and Biomarkers of Response
Brief Title: Intensity Modulated Radiation Therapy (IMRT) for Patients With Rectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed to enrollment due to slow accrual.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-157
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Rectal Cancer
Keywords: IMRT; radiation therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Short course IMRT (Experimental): Patients will receive short course IMRT (Intensity Modulated Radiation Therapy) prior to surgery. Dose will be 5 Gy x 5, followed by surgery the week after
  Interventions: Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy — Radiation therapy once a day for 5 days
  Other Names: IMRT

SUMMARY:
This study will investigate short course radiation therapy using IMRT as an alternative to standard chemo radiation because prior studies have shown that this method of treatment will potentially reduce some fo the side effects of standard treatment, improve quality of life, and help to control the growth of rectal cancer cells. IMRT is a type of radiation that uses computer-generated images to match radiation to the size and shape of the tumor. Since the intensity of each radiation beam can be controlled, the radiation dose can wrap around normal tissue which allows the study doctor to deliver a higher dose of radiation to the tumor with less damage to nearby healthy tissue. The purpose of this research study is to see what impact this treatment will have on quality of life, as well as to see if there are any late side effects that come about after the participant has completed the treatment.

DETAILED DESCRIPTION:
* Radiation treatment to the rectum will be given once a day, for 5 days. Each radiation treatment will take about 20-30 minutes.
* The following procedures will be performed on day 1 of radiation treatment: physical examination, blood tests and quality of life questionnaire.
* During radiation treatment a physical examination will be performed once during the 5 days of radiation treatment. A Quality of Life Questionnaire will be administered on the last day of radiation treatment.
* Surgery will be performed within 3-14 days after the last day of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the rectum
* T3 or N+ disease by MRI or endoscopic ultrasound. Metastatic disease is permitted, except for known brain metastases, as long as local treatment with RT and surgery is recommended.
* Prior chemotherapy is permitted. For patients who have previously received bevacizumab, the last dose must be greater than 4 weeks prior to initiation of radiation therapy.
* 18 years of age or older
* Life expectancy of greater than 3 months
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0, 1 or 2
* Normal organ and marrow function as outlined in the protocol
* Women of child-bearing potential and men must agree to use of adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Pelvic radiotherapy prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Participants may not be receiving any other investigational agents. Patients may not be receiving any other treatment for their rectal cancer during study participation
* Participants with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of known radiation sensitivity syndrome
* History of inflammatory bowel disease
* Active scleroderma or CREST syndrome
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S. Hong, MD, Principal Investigator — Massachusetts General Hosptial
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Short Course IMRT: Pts will receive short course IMRT prior to surgery. Dose will be 5 Gy x 5, followed by surgery the week after
  Intensity Modulated Radiation Therapy: Radiation therapy once a day for 5 days
Period: Overall Study
Arm/Group | Short Course IMRT
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Short Course IMRT
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Bowel Quality of Life
Description: To determine the rate of fecal incontinence at 1 year in patients undergoing an low anterior resection (LAR), as measured by bowel quality of life measure after preoperative conformal radiation therapy delivered in one week for rectal cancer.
Time Frame: 2 years
Population: Study was terminated early due to slow accrual. Analysis was not performed.
Arm/Group | Short Course IMRT
Number analyzed (Participants) | 0

2. Secondary Outcome: Pelvic Control Rate
Description: To determine the pelvic control rate of patients after short course radiation therapy and surgery.
Time Frame: 2 years
Population: Study was closed early due to poor accrual. Analyses not completed.
Arm/Group | Short Course IMRT
Number analyzed (Participants) | 0

3. Secondary Outcome: Surgical Complication Rate
Description: To determine the surgical complication rate in patients who received preoperative radiation therapy.
Time Frame: 2 years
Population: Study was closed early due to poor accrual. Analyses not completed.
Arm/Group | Short Course IMRT
Number analyzed (Participants) | 0

4. Secondary Outcome: Tissue Microarray
Description: To determine changes in the tumor induced by radiation as assessed by tissue microarray.
Time Frame: 2 years
Population: Study was closed early due to poor accrual. Analyses not completed.
Arm/Group | Short Course IMRT
Number analyzed (Participants) | 0

5. Secondary Outcome: Quantity of Circulating Tumor Cells
Description: To determine the impact of radiation and surgery on quantity of circulating tumor cells in both metastatic and non-metastatic patients.
Time Frame: 2 years
Population: Study was closed early due to poor accrual. Analyses not completed.
Arm/Group | Short Course IMRT
Number analyzed (Participants) | 0

6. Secondary Outcome: Accuracy
Description: To determine the accuracy of advanced MRI imaging and PET (Positron Electron Tomography) /CT in predicting nodal stage.
Time Frame: 2 years
Population: Study was closed early due to poor accrual. Analyses not completed.
Arm/Group | Short Course IMRT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 Days
Description: Adverse events experienced by participants will be collected and reported from initiation of study treatment, throughout the study, and within 30 days of the last dose of study treatment.
Arm/Group | Short Course IMRT
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Short Course IMRT (N=2)
urinary tract infection (Infections and infestations) | 1
vomiting (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 1
confusion (Nervous system disorders) | 1
urinary retention (Renal and urinary disorders) | 1
platelets (Blood and lymphatic system disorders) | 1
elevated bilirubin (Metabolism and nutrition disorders) | 1
low phosphorus (Metabolism and nutrition disorders) | 1
anemia (Blood and lymphatic system disorders) | 1
fever (General disorders) | 1
cellulitis (Skin and subcutaneous tissue disorders) | 1
lymphopenia (Blood and lymphatic system disorders) | 2
leukopenia (Blood and lymphatic system disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 2
diarrhea (Gastrointestinal disorders) | 1
edema (Blood and lymphatic system disorders) | 1 — lower extremity
erythema (Skin and subcutaneous tissue disorders) | 1
pilonidal abscess (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Study was closed early due to poor accrual. Analyses not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No